CLINICAL TRIAL: NCT02889120
Title: Telemedicine Performed by General Practitioners in Medical Call Centres:Quality Assessment of Drug Prescription by Phone
Brief Title: Assessment of Drug Prescription by Phone
Acronym: TELEPRES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Nantes University Hospital (Other); Central Hospital, Nancy, France (Other); Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/197
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Drug Advice by Phone
Keywords: Drug advice by phone; Teleprescription; Medical call centre; Out of hours call

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prescription of medicines by telephone in French medical call Centres is a part of the general practitioners activity.

This study aimed to described drug prescription by phone (MTP) performed in four medical call centers. The primary objective is to evaluate adherence to french practice guidelines for the drug prescription by phone (Haute Autorité de Santé, 2009) The secondary objective is to evaluate the risk/benefit ratio for drug prescription by phone.

ELIGIBILITY:
Inclusion Criteria:

* All phone calls, from september to october 2013, leading to a drug prescription by a general practitioner of four medical call centres..

Exclusion Criteria:

* Medical emergency
* Patient refusing or not able to provide consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All phone calls, from september to october 2013, leading to a drug prescription by a general practitioner of four medical call centres were eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1263 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Adherence to Practice Guidelines for the drug prescription by phone | 3 days
  The aim is to measure the adherence to HAS (Haute Autorité de Santé, 2009) pratice guidelines for the drug prescription by phone
Risk/benefit ratio for drug prescription by phone | 3 days

IPD SHARING:
Plan to Share IPD: No